CLINICAL TRIAL: NCT00931892
Title: Circulating Markers of Celiac Disease Activity During Gluten Challenge - a Pilot Study.
Brief Title: Serum Markers in Gluten Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ciaran Kelly, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007P000280; K23DK082619 (NIH)
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Results first posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Celiac Disease
Keywords: celiac disease; gluten challenge
MeSH Terms: conditions — Celiac Disease | interventions — Glutens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low gluten group (Experimental): Subjects will eat 3g of gluten per day
  Interventions: Dietary Supplement: Gluten
- High gluten group (Experimental): Subjects will eat 10g of gluten per day
  Interventions: Dietary Supplement: Gluten

INTERVENTIONS:
Dietary Supplement: Gluten — 3g
  Arms: Low gluten group
Dietary Supplement: Gluten — 10g
  Arms: High gluten group

SUMMARY:
1. The purpose of this research study is to evaluate non-invasive markers of celiac disease activity in subjects that are on a gluten-free diet, in remission from celiac disease who undergo gluten challenge.
2. The secondary aims of this protocol are to identify novel mediators important in the pathophysiology of celiac disease and to evaluate changes in metabolism with gluten exposure.

DETAILED DESCRIPTION:
The diagnosis of celiac disease carries with it important ramifications. Celiac disease is a systemic immunologic disorder in which the sentinel lesion is an enteropathy triggered by polypeptides derived primarily from the gliadin proteins found in wheat, rye and barley. Ingestion of the offending proteins leads to inflammation and intestinal mucosal damage, which results in a spectrum of abdominal symptoms, increased intestinal permeability, malabsorption, occult gastrointestinal bleeding and diarrhea. Systemic manifestations of celiac disease include a myriad of conditions including malignancy and autoimmune disease.

The only accepted treatment for celiac disease is lifelong adherence to a gluten free diet. Adherence to this diet, simply put avoiding all foods containing even small amounts of wheat, rye and barley, has been shown to lead to improvement in the majority of related problems and normalization of all standard diagnostic tests. Because of this many individuals who present for evaluation of possible celiac disease but who are already on a gluten free diet cannot be tested accurately as there is currently no way of differentiating between healthy individuals and individuals with well treated celiac disease. The standard practice in such cases is to perform a 'Gluten Challenge' whereby the patient eats the equivalent of 2 slices of bread per day for six to eight weeks before returning for evaluation with serologic testing and endoscopy with duodenal biopsy. The use of the gluten challenge in clinical practice is limited by patient symptoms and resistance to such a long test period, after which it may take a number of weeks for the intestine to heal and the symptoms to resolve. Autoantibodies to tissue transglutaminase or antibodies to deamidated gliadin, while being excellent tools to predict celiac disease in patients who have been on a long-term gluten containing diet, display low sensitivities to detect short-term and/or recent gluten exposure. For this reason, it would be very useful if novel circulating markers could be identified that indicate the presence of celiac disease and in particular would provide an early and less invasive marker of a positive response to gluten challenge.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 17 and 72 years, inclusive.
2. Subject must have been diagnosed with celiac disease by duodenal / jejunal biopsy at least 6 months prior to entrance into the study.
3. Subject has Anti-Tissue Transglutaminase (anti-tTG) ≤ 20 EU as measured by serology.
4. Subject must be on a gluten-free diet for at least the past 6 months.
5. Female subjects should be either post-menopausal (amenorrhea for at least 24 consecutive months), surgically sterile, or women of child-bearing potential (WOCP) with a negative urine beta human chorionic gonadotropin (HCG) pregnancy test prior to entering the study and who are using or agree to use acceptable methods of contraception. Abstinence is an acceptable means of avoiding pregnancy as long as the subject agrees to use contraception if they become sexually active. Acceptable contraceptives include intrauterine devices (IUDs), hormonal contraceptives (oral, depo, patch or injectable) in use for one month prior to screening and double barrier methods such as condoms or diaphragms with spermicidal gel or foam.
6. Subject must sign an Institutional Review Board approved informed consent and agree to complete required clinic visits.
7. BMI between 18.5 and 38, inclusive.

Exclusion Criteria:

1. Subject has Anti-Tissue Transglutaminase (anti-tTG) > 20 EU as measured by serology.
2. Subject has other food intolerances or food allergies (other than celiac disease) that would interfere with the conduct of the study).
3. Subject has a history of severe acute symptomatic reactions to sporadic gluten ingestion
4. Subject has any chronic active GI disease other than celiac disease (e.g. Crohn's disease, IBS).
5. Subjects with symptomatic neurological or psychiatric disease(s) that would interfere with the conduct of the study.
6. Subject has clinically significant abnormal laboratory test results at the screening visit or as determined by the Principal Investigator
7. Subject is pregnant or breast feeding.
8. Subject (premenopausal females) is sexually active without contraception.
9. Subject should not have been on steroids in the past 3 months.
10. Subject is deemed inappropriate by the Principal Investigator.

Ages: 17 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ciaran P Kelly, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Daniel A Leffler, MD, MS, Study Director — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Svedlund J, Sjodin I, Dotevall G. GSRS--a clinical rating scale for gastrointestinal symptoms in patients with irritable bowel syndrome and peptic ulcer disease. Dig Dis Sci. 1988 Feb;33(2):129-34. doi: 10.1007/BF01535722. PMID 3123181
- [Result] Adelman DC, Murray J, Wu TT, Maki M, Green PH, Kelly CP. Measuring Change In Small Intestinal Histology In Patients With Celiac Disease. Am J Gastroenterol. 2018 Mar;113(3):339-347. doi: 10.1038/ajg.2017.480. Epub 2018 Feb 20. PMID 29460921
- [Result] Leffler DA, Dennis M, Edwards George J, Jamma S, Cook EF, Schuppan D, Kelly CP. A validated disease-specific symptom index for adults with celiac disease. Clin Gastroenterol Hepatol. 2009 Dec;7(12):1328-34, 1334.e1-3. doi: 10.1016/j.cgh.2009.07.031. Epub 2009 Aug 7. PMID 19665584
- [Derived] Leffler D, Schuppan D, Pallav K, Najarian R, Goldsmith JD, Hansen J, Kabbani T, Dennis M, Kelly CP. Kinetics of the histological, serological and symptomatic responses to gluten challenge in adults with coeliac disease. Gut. 2013 Jul;62(7):996-1004. doi: 10.1136/gutjnl-2012-302196. Epub 2012 May 22. PMID 22619366
- See also: BIDMC Celiac Center Research website — http://www.bidmc.org/CentersandDepartments/Departments/DigestiveDiseaseCenter/CeliacDiseaseCenter/ResearchStudies.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 21 patients were enrolled in the study. 1 patient was found to be negative for DQ2 and DQ8, therefore did not have Celiac disease. This patient was excluded from the study. Therefore, for the study we had a total of 20 participants.
Period: Completed Gluten Challenge
Arm/Group | Low Gluten Group | High Gluten Group
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Completed Endoscopies
Arm/Group | Low Gluten Group | High Gluten Group
Started | 10 | 10
First Endoscopy | 10 | 10
Second Endoscopy | 10 | 10
Third Endoscopy | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Patient did not complete third endoscopy due to discomfort | 0 | 1

BASELINE CHARACTERISTICS:
Population: Subjects with biopsy proven coelic dieasese in remission were enrolled.
Groups:
- Low Gluten Group: Participants meeting inclusion criteria were randomized into the low gluten group. These participants ate two slices of wheat bread per day (3 g of gluten). Bread was procured from a standard source and gluten dose tested using the RIDASCREEN Gliadin R5 antibody ELISA. The study included a 14-day run-in period followed by a 14 day gluten challenge and a final visit 14 days post-gluten challenge. Other than the dispensed bread, subjects were instructed to remain on their gluten-free diet throughout the duration of the study.
  Gluten: 3g
- High Gluten Group: Participants meeting inclusion criteria were randomized into the low gluten group. These participants ate five slices of wheat bread per day (10 g of gluten). Bread was procured from a standard source and gluten dose tested using the RIDASCREEN Gliadin R5 antibody ELISA. The study included a 14-day run-in period followed by a 14 day gluten challenge and a final visit 14 days post-gluten challenge. Other than the dispensed bread, subjects were instructed to remain on their gluten-free diet throughout the duration of the study.
  Gluten: 10g
- Total: Total of all reporting groups
Arm/Group | Low Gluten Group | High Gluten Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (13.0) | 38.8 (13.1) | 43.3 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Age at Celiac Diagnosis [Mean (Standard Deviation); unit: years] | 45.4 (13.9) | 31.0 (11.7) | 35.7 (14.4)
Months since Celiac Disease diagnosis [Mean (Standard Deviation); unit: months] | 42.3 (21.3) | 92.5 (49.1) | 62.3 (87.1)
Laboratory Characteristics [Count of Participants; unit: Participants]
  HLA DQ2 | 4 | 6 | 10
  HLA DQ8 | 3 | 3 | 6
  HLA DQ2 + DQ 8 | 1 | 1 | 2
  HLA A1 * 05 alone | 2 | 0 | 2
Villous height to crypt depth ratio [Mean (Standard Deviation); unit: unitless] — Villous height to crypt depth (Vh: Cd) ratio was determined by measuring the mean height/mean depth of adjacent villi/proliferative crypt zones at magnification 100x
  Vh:Cd and IEL count Adelman DC, Murray J, Wu TT, Mäki M, Green PH, Kelly CP. Measuring Change In Small Intestinal Histology In Patients With Celiac Disease. Am J Gastroenterol. 2018 Mar;113(3):339-347. doi: 10.1038/ajg.2017.480. Epub 2018 Feb 20. Review. PubMed PMID: 29460921.
  unitless | 2.05 (0.80) | 4.33 (6.69) | 2.21 (0.8)
Mean number of Intraepithelial lymphocytes [Mean (Standard Deviation); unit: unitless] — Villous lymphocyte infiltration was recorded at magnification 300 x as number of intraepithelial lymphocytes (IEL count) per 100 enterocytes
  Vh:Cd and IEL count Adelman DC, Murray J, Wu TT, Mäki M, Green PH, Kelly CP. Measuring Change In Small Intestinal Histology In Patients With Celiac Disease. Am J Gastroenterol. 2018 Mar;113(3):339-347. doi: 10.1038/ajg.2017.480. Epub 2018 Feb 20. Review. PubMed PMID: 29460921.
  unitless | 37.10 (13.66) | 28.4 (13.3) | 32.59 (15.1)
Baseline tissue transglutaminase (tTG) [Mean (Standard Deviation); unit: units] — NEGATIVE <20, BORDERLINE 20-30, POSITIVE >30
  units | 13.76 (8.30) | 8.27 (5.70) | 11.00 (7.50)
Baseline Deamidated gliadin peptide (DGP) [Mean (Standard Deviation); unit: units] — NEGATIVE <20, BORDERLINE 20-30, POSITIVE >30 METHOD IS INOVA ANTI-DEAMIDATED GLIADIN PEPTIDE IGA/IGG.
  units | 6.70 (2.59) | 14.04 (26.49) | 10.90 (19.60)
Baseline Celiac Dietary Adherence test (CDAT) [Mean (Standard Deviation); unit: scores on a scale] — CDAT scores range from 7-35 for scores. Lower scores indicate better dietary adherence
  scores on a scale | 11.33 (3.2) | 11.40 (2.9) | 11.37 (2.9)
Baseline Celiac Symptom Index (CSI) [Mean (Standard Deviation); unit: scores on a scale] — CSI (Celiac Symptom Index) scores range from 7-80. Higher scores indicate greater degree of symptoms
  CSI:
  Leffler DA, Dennis M, Edwards George J, Jamma S, Cook EF, Schuppan D, Kelly CP. A validated disease-specific symptom index for adults with celiac disease. Clin Gastroenterol Hepatol. 2009;7:1328-34. PubMed PMID: 19665584.
  scores on a scale | 28.50 (5.78) | 22.50 (4.99) | 25.26 (5.90)
Baseline Gastrointestinal Symptom Rating Scale (GSRS) [Mean (Standard Deviation); unit: scores on a scale] — GSRS (Gastrointestinal Symptom Rating Scale) scores range 15-105 with higher scores indicating greater degree of symptoms
  GSRS:
  Svedlund J, Sjödin I, Dotevall G. GSRS--a clinical rating scale for gastrointestinal symptoms in patients with irritable bowel syndrome and peptic ulcer disease. Dig Dis Sci. 1988;33(2):129-134. doi:10.1007/BF01535722
  scores on a scale | 22.88 (9.58) | 19.20 (3.26) | 20.32 (5.10)
Baseline Quality of Life Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: scores on a scale] — VAS (Quality of Life Visual Analog Scale) scores range from 0-100 with higher scores indicating better health related quality of life
  scores on a scale | 80.00 (13.10) | 84.40 (12.10) | 82.20 (12.50)

OUTCOME MEASURES:

1. Primary Outcome: Crypt Depth to Villous Height Ratio
Description: Histological evaluation of duodenal biopsy samples to evaluate crypt depth to villous height ratio. On the best oriented section of each biopsy fragment, villous height to crypt depth (Vh:Cd) ratio was determined by measuring the mean height /mean depth of adjacent villi/proliferative crypt zones at magnification 100x. Evaluations were considered discrepant Vh:Cd differed by more than 0.5. Overall, there was excellent concordance with the evaluations of the 165 biopsy fragments determined to be optimal for evaluation.
  The Vh:Cd ratios on individual biopsies from a single averaged to produce a representative Vh:Cd ratio for each endoscopy. Normal Vh:Cd ratio was regarded as 3:1 or greater.
  Adelman DC, Murray J, Wu TT, Mäki M, Green PH, Kelly CP. Measuring Change In Small Intestinal Histology In Patients With Celiac Disease. Am J Gastroenterol. 2018 Mar;113(3):339-347. doi: 10.1038/ajg.2017.480. Epub 2018 Feb 20. Review. PubMed PMID: 29460921.
Time Frame: Screening (Day -7 to -14), Day 3, Day 14
Population: Subjects with biopsy proven celiac disease in remission were enrolled. For Day 3, 17 subjects had evaluable pathology biopsies. On Day 14, 19 participants had evaluable pathology biopsies.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Baseline (Day -14) Low Gluten Group; Day 3 Low Gluten Group; Day 14 Low Gluten Group: Villous height to crypt depth ratio in low gluten group
  In the low gluten group, subjects consumed 3 grams of gluten per day
- Baseline (Day -14) High Gluten Group; Day 3 High Gluten Group: Villous height to crypt depth ratio in high gluten group
  In the high gluten group, subjects consumed 10 grams of gluten per day.
- Day 14 High Gluten Group: Villous height to crypt depth ratio in high gluten group.
  In the high gluten group subjects consume 10 grams of gluten per day.
Arm/Group | Baseline (Day -14) Low Gluten Group | Baseline (Day -14) High Gluten Group | Day 3 Low Gluten Group | Day 3 High Gluten Group | Day 14 Low Gluten Group | Day 14 High Gluten Group
Number analyzed (Participants) | 10 | 10 | 8 | 9 | 10 | 9
ratio | 2.05 (0.80) | 4.33 (6.69) | 1.19 (0.67) | 2.02 (0.99) | 0.98 (0.85) | 1.26 (1.08)
Statistical Analysis 1: Comparison: Baseline (Day -14) Low Gluten Group vs Baseline (Day -14) High Gluten Group vs Day 3 Low Gluten Group vs Day 3 High Gluten Group vs Day 14 Low Gluten Group vs Day 14 High Gluten Group; Test type: Other; p = 0.670, t-test, 2 sided

2. Secondary Outcome: Count of Intraepithelial Lymphocytes Per 100 Enterocytes in Duodenal Biopsy Samples
Description: On the best oriented section of each biopsy fragment , the number of intraepithelial lymphocytes (IEL count) per 100 enterocytes was recorded at magnification 400x. IEL counts were considered discrepant if a difference of >10 IELs existed between counts. Overall, there was excellent concordance with the evaluations of the 165 biopsy fragments determined to be optimal for evaluation.
  The IEL counts on individual biopsies from a single endoscopy were averaged to produce a representative IEL count for each endoscopy.
  Adelman DC, Murray J, Wu TT, Mäki M, Green PH, Kelly CP. Measuring Change In Small Intestinal Histology In Patients With Celiac Disease. Am J Gastroenterol. 2018 Mar;113(3):339-347. doi: 10.1038/ajg.2017.480. Epub 2018 Feb 20. Review. PubMed PMID: 29460921.
Time Frame: Screening (Day -7 to -14), Day 3, Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Count of Lymphocytes Per 100 Enterocytes
Groups:
- Baseline (Day -14) Low Gluten Dose Group; Day 3 Low Gluten Dose Group; Day 14 Low Gluten Dose Group: Intraepithelial lymphocyte count(per 100 enterocytes) in low gluten dose groups.
  Subjects in the low gluten dose group consumed 3 grams of gluten per day.
- Baseline (Day -14) High Gluten Dose Group; Day 14 High Gluten Dose Group: Intraepithelial lymphocyte count(per 100 enterocytes) in high gluten dose groups.
  Subjects in the high gluten dose group consumed 10 grams of gluten per day
- Day 3 High Gluten Dose Group: Intraepithelial lymphocyte count(per 100 enterocytes) in high gluten dose groups.
  Subjects in the low gluten dose group consumed 10 grams of gluten per day
Arm/Group | Baseline (Day -14) Low Gluten Dose Group | Baseline (Day -14) High Gluten Dose Group | Day 3 Low Gluten Dose Group | Day 3 High Gluten Dose Group | Day 14 Low Gluten Dose Group | Day 14 High Gluten Dose Group
Number analyzed (Participants) | 10 | 10 | 8 | 9 | 10 | 9
Count of Lymphocytes Per 100 Enterocytes | 37.08 (13.66) | 28.91 (15.81) | 44.89 (20.49) | 30.68 (18.09) | 47.95 (14.30) | 52.36 (28.52)
Statistical Analysis 1: Comparison: Baseline (Day -14) Low Gluten Dose Group vs Baseline (Day -14) High Gluten Dose Group vs Day 3 Low Gluten Dose Group vs Day 3 High Gluten Dose Group vs Day 14 Low Gluten Dose Group vs Day 14 High Gluten Dose Group; Test type: Other; p = 0.409, t-test, 2 sided

3. Secondary Outcome: Measures of Intestinal Permeability (Urinary Lactulose to Mannitol Ratio)
Description: LAMA evaluation has been reported to be an accurate measure of small intestinal mucosal permeability though assessment of differential absorption of lactulose and mannitol. For LAMA testing, a solution containing 7.5 g lactulose and 2 g mannitol in 100 mL of water was ingested by the participants in the evening after visit 1 and in the evening before each other study visit. The participants were asked to fast for at least 4 h and to void completely before drinking the sugar solution, then fast overnight and collect all overnight and morning urine. Urine sample analyzed for lactulose and mannitol using standardized methodology by liquid chromatography-tandem mass spectrometry.
Time Frame: Screening (Day -7 to -14), Day 0, Day 3, Day 7, Day 14, Day 28
Population: Subjects with biopsy proven celiac disease in remission were enrolled. Measures of intestinal permeability (urinary lactulose to mannitol ratio) (LAMA) . Four participants were unable to tolerate LAMA testing due to gastrointestinal symptoms.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Day -14 Low Gluten Dose Group; Day 0 Low Gluten Dose Group; Day 3 Low Gluten Dose Group; Day 7 Low Gluten Dose Group; Day 14 Low Gluten Dose Group; Day 28 Low Gluten Dose Group: Subjects in the low gluten dose group consumed 3 grams of gluten per day.
- Day -14 High Gluten Dose Group; Day 0 High Gluten Dose Group; Day 3 High Gluten Dose Group; Day 7 High Gluten Dose Group; Day 14 High Gluten Dose Group; Day 28 High Gluten Dose Group: Subjects in the high gluten dose group consumed 10 grams of gluten per day.
Arm/Group | Day -14 Low Gluten Dose Group | Day -14 High Gluten Dose Group | Day 0 Low Gluten Dose Group | Day 0 High Gluten Dose Group | Day 3 Low Gluten Dose Group | Day 3 High Gluten Dose Group | Day 7 Low Gluten Dose Group | Day 7 High Gluten Dose Group | Day 14 Low Gluten Dose Group | Day 14 High Gluten Dose Group | Day 28 Low Gluten Dose Group | Day 28 High Gluten Dose Group
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 7 | 8 | 7 | 8 | 6 | 8 | 7
ratio | 0.23 (0.17) | 0.24 (0.25) | 0.65 (1.15) | 0.17 (0.15) | 0.25 (0.15) | 0.44 (0.60) | 0.45 (0.71) | 0.29 (0.28) | 0.89 (1.53) | 0.59 (0.52) | 0.29 (0.24) | 0.57 (0.82)
Statistical Analysis 1: Comparison: Day 14 Low Gluten Dose Group vs Day 14 High Gluten Dose Group vs Day 28 Low Gluten Dose Group vs Day 28 High Gluten Dose Group; Test type: Other; p = 0.387, t-test, 2 sided
Statistical Analysis 2: Comparison: Day 0 Low Gluten Dose Group vs Day 0 High Gluten Dose Group vs Day 28 Low Gluten Dose Group vs Day 28 High Gluten Dose Group; Test type: Other; p = 0.208, t-test, 2 sided

4. Secondary Outcome: Measures of Immune Activation
Description: IgA anti-human tissue transglutaminase assay (Inova Diagnostics, Inc., San Diego, USA): negative <20, borderline 20-30, positive >30.
  IgA/IgG anti- DGP assay : NEGATIVE <20, BORDERLINE 20-30, POSITIVE >30 METHOD IS INOVA ANTI-DEAMIDATED GLIADIN PEPTIDE IGA/IGG.
Time Frame: Screening (Day -7 to -14), Day 0, Day 3, Day 7, Day 14, Day 28
Population: Subjects with biopsy proven celiac disease in remission were enrolled.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Day -14 Low Gluten Dose Group | Day -14 High Gluten Dose Group | Day 0 Low Gluten Dose Group | Day 0 High Gluten Dose Group | Day 3 Low Gluten Dose Group | Day 3 High Gluten Dose Group | Day 7 Low Gluten Dose Group | Day 7 High Gluten Dose Group | Day 14 Low Gluten Dose Group | Day 14 High Gluten Dose Group | Day 28 Low Gluten Dose Group | Day 28 High Gluten Dose Group
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
units on a scale
  IgA anti-tTG | 6.70 (2.60) | 10.34 (5.75) | 13.76 (10.88) | 11.50 (6.63) | 11.84 (9.50) | 10.34 (5.75) | 13.77 (10.90) | 11.50 (6.63) | 12.63 (8.73) | 15.16 (10.30) | 37.81 (45.07) | 43.20 (53.77)
  IgA/IgG anti- DGP | 6.70 (2.60) | 14.04 (26.49) | 7.83 (2.54) | 14.69 (27.01) | 12.95 (8.26) | 14.04 (26.49) | 7.83 (2.54) | 14.69 (27.01) | 17.81 (22.97) | 22.74 (29.31) | 45.42 (62.56) | 41.95 (33.91)
Statistical Analysis 1: Comparison: Day -14 Low Gluten Dose Group vs Day -14 High Gluten Dose Group vs Day 14 Low Gluten Dose Group vs Day 14 High Gluten Dose Group; P Value for IgA anti-tTG; Test type: Superiority; p = 0.010, ANOVA
Statistical Analysis 2: Comparison: Day -14 Low Gluten Dose Group vs Day -14 High Gluten Dose Group vs Day 14 Low Gluten Dose Group vs Day 14 High Gluten Dose Group; P Value for IgA/IgG anti-DGP; Test type: Superiority; p = 0.036, ANOVA
Statistical Analysis 3: Comparison: Day -14 Low Gluten Dose Group vs Day -14 High Gluten Dose Group vs Day 28 Low Gluten Dose Group vs Day 28 High Gluten Dose Group; P Value for IgA anti-tTG; Test type: Superiority; p = 0.013, ANOVA
Statistical Analysis 4: Comparison: Day -14 Low Gluten Dose Group vs Day -14 High Gluten Dose Group vs Day 28 Low Gluten Dose Group vs Day 28 High Gluten Dose Group; P Value for IgA/IgG anti-DGP; Test type: Superiority; p = 0.006, ANOVA

5. Secondary Outcome: Assessment of Protein Expression in Intestinal Biopsies
Description: Proportion of participants responding to a gluten challenge. Tissue transglutaminase (tTG) scoring: NEGATIVE <20, BORDERLINE 20-30, POSITIVE >30. Deamidated gliadin peptide (DGP) scoring: NEGATIVE <20, BORDERLINE 20-30, POSITIVE >30 METHOD IS INOVA ANTI-DEAMIDATED GLIADIN PEPTIDE IGA/IGG.
Time Frame: Screening (Day -7 to -14), Day 3, Day 14
Population: All 20 subjects were included for the tTG and DGP analysis. For Day 28 High Gluten Challenge Dose Group, 1 participant had both a tTG and DGP >20 which is why the count is greater than the number analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Day 14 High Gluten Challenge Group; Day 28 High Gluten Dose Group; Day 14 or Day 28 High Gluten Dose Group: Subjects in the high gluten dose group consumed 10 grams of gluten per day
- Day 14 or Day 28 Low Gluten Dose Group: Subjects in the low gluten dose group consumed 3 grams of gluten per day
Arm/Group | Day 14 Low Gluten Dose Group | Day 14 High Gluten Challenge Group | Day 28 Low Gluten Dose Group | Day 28 High Gluten Dose Group | Day 14 or Day 28 Low Gluten Dose Group | Day 14 or Day 28 High Gluten Dose Group
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 20 | 20
Participants
  tTG > 20 | 3 | 2 | 5 | 6 | 8 | 8
  DGP > 20 | 2 | 4 | 4 | 5 | 6 | 9
  tTG > 20 or DGP > 20 | 5 | 6 | 9 | 10 | 14 | 17

6. Secondary Outcome: Symptomatic Response to Gluten Exposure Determined by Celiac Symptom Index Questionnaire
Description: CSI (Celiac Symptom Index) scores range from 7-80. Higher scores indicate greater degree of symptoms
  CSI:
  Leffler DA, Dennis M, Edwards George J, Jamma S, Cook EF, Schuppan D, Kelly CP. A validated disease-specific symptom index for adults with celiac disease. Clin Gastroenterol Hepatol. 2009;7:1328-34. PubMed PMID: 19665584.
Time Frame: Screening (Day -7 to -14), Day 0, Day 3, Day 7, Day 14, Day 28
Population: Subjects with biopsy proven celiac disease in remission were enrolled. On Day -14, one subject in the high gluten dose group missed the CSI. On Day 7 one subject in the high gluten dose group missed the CSI. On Day 14 one subject in the high gluten dose group missed the CSI. On Day 28, one subject in the high gluten dose group and one subject in the low gluten dose missed the CSI.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Day -14 Low Gluten Dose Group | Day -14 High Gluten Dose Group | Day 0 Low Gluten Dose Group | Day 0 High Gluten Dose Group | Day 3 Low Gluten Dose Group | Day 3 High Gluten Dose Group | Day 7 Low Gluten Dose Group | Day 7 High Gluten Dose Group | Day 14 Low Gluten Dose Group | Day 14 High Gluten Dose Group | Day 28 Low Gluten Dose Group | Day 28 High Gluten Dose Group
Number analyzed (Participants) | 10 | 9 | 10 | 10 | 10 | 10 | 10 | 9 | 10 | 9 | 9 | 9
score on a scale | 28.5 (5.78) | 22.5 (4.99) | 28.44 (6.44) | 23.00 (5.29) | 30.33 (7.81) | 27.54 (10.27) | 31.11 (7.90) | 28.80 (13.36) | 31.38 (11.40) | 31.00 (12.70) | 26.88 (7.70) | 23.90 (6.740)
Statistical Analysis 1: Comparison: Day 3 Low Gluten Dose Group vs Day 3 High Gluten Dose Group; P Value for Celiac Symptom Index (CSI) score for Day 3 of Gluten Challenge; Test type: Other; p = 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Day -14 Low Gluten Dose Group vs Day -14 High Gluten Dose Group vs Day 14 Low Gluten Dose Group vs Day 14 High Gluten Dose Group; P Value for Celiac Symptom Index (CSI) Score from baseline to Day 14; Test type: Other; p = 0.020, t-test, 2 sided
Statistical Analysis 3: Comparison: Day -14 Low Gluten Dose Group vs Day -14 High Gluten Dose Group vs Day 0 Low Gluten Dose Group vs Day 0 High Gluten Dose Group vs Day 3 Low Gluten Dose Group vs Day 3 High Gluten Dose Group vs Day 7 Low Gluten Dose Group vs Day 7 High Gluten Dose Group vs Day 14 Low Gluten Dose Group vs Day 14 High Gluten Dose Group vs Day 28 Low Gluten Dose Group vs Day 28 High Gluten Dose Group; P Value for Celiac Symptom Index (CSI)score between high gluten group and low gluten group across study; Test type: Superiority; p = 0.060, ANOVA

7. Secondary Outcome: Assessment of Protein Expression in Intestinal Biopsies Using Marsh Scores
Description: as for outcome 5
Time Frame: Screening (Day -7 to -14), Day 3, Day 14
Population: Only 19 subjects were evaluated for Marsh scores because one patient had a single endoscopy which did not produce evaluable samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Day 14 Low Gluten Dose Group | Day 14 High Gluten Challenge Group | Day 28 Low Gluten Dose Group | Day 28 High Gluten Dose Group | Day 14 or Day 28 Low Gluten Dose Group | Day 14 or Day 28 High Gluten Dose Group
Number analyzed (Participants) | 10 | 9 | 10 | 9 | 20 | 19
Participants
  Marsh III | 5 | 8 | 0 | 0 | 5 | 8
  Marsh III or tTG >20 | 8 | 9 | 5 | 6 | 13 | 16
  Marsh III or DGP > 20 | 7 | 9 | 4 | 5 | 11 | 17
  Marsh III or DGP > 20 or tTG > 20 | 10 | 9 | 9 | 9 | 19 | 19

8. Secondary Outcome: Symptomatic Response to Gluten Exposure Determined by Gastrointestinal Symptom Rating Scale
Description: Measure Description: GSRS (Gastrointestinal Symptom Rating Scale) scores range 15-105 with higher scores indicating greater degree of symptoms
  GSRS:
  Svedlund J, Sjödin I, Dotevall G. GSRS--a clinical rating scale for gastrointestinal symptoms in patients with irritable bowel syndrome and peptic ulcer disease. Dig Dis Sci. 1988;33(2):129-134. doi:10.1007/BF01535722
Time Frame: Screening (Day -7 to -14), Day 0, Day 3, Day 7, Day 14, Day 28
Population: Subjects with biopsy proven celiac disease in remission were enrolled. On Day -14, one subject in the high gluten group missed completing the GSRS. On Day 0, two subjects (one in the low gluten group and one subject in the high gluten group) missed completing the GSRS. On Day 7, one subject in the high gluten group missed completing the GSRS. On Day 14, one subject in the high gluten group missed completing the GSRS. On Day 28, one subject in the high gluten group missed completing the GSRS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Day -14 Low Gluten Dose Group | Day -14 High Gluten Dose Group | Day 0 Low Gluten Dose Group | Day 0 High Gluten Dose Group | Day 3 Low Gluten Dose Group | Day 3 High Gluten Dose Group | Day 7 Low Gluten Dose Group | Day 7 High Gluten Dose Group | Day 14 Low Gluten Dose Group | Day 14 High Gluten Dose Group | Day 28 Low Gluten Dose Group | Day 28 High Gluten Dose Group
Number analyzed (Participants) | 10 | 9 | 9 | 9 | 10 | 10 | 10 | 9 | 10 | 9 | 10 | 9
score on a scale | 21.63 (7.05) | 19.20 (3.26) | 22.88 (9.58) | 18.40 (3.06) | 30.22 (11.63) | 26.45 (13.18) | 28.22 (9.87) | 27.30 (14.94) | 31.00 (13.71) | 31.00 (17.09) | 23.89 (11.59) | 19.40 (4.33)
Statistical Analysis 1: Comparison: Day 3 Low Gluten Dose Group vs Day 3 High Gluten Dose Group; P Value for the Gastrointestinal Symptom Rating Scale (GSRS) on Day 3 of the Gluten Challenge; Test type: Other; p = 0.01, t-test, 2 sided
Statistical Analysis 2: Comparison: Day -14 Low Gluten Dose Group vs Day -14 High Gluten Dose Group vs Day 14 Low Gluten Dose Group vs Day 14 High Gluten Dose Group; P Value for Gastrointestinal Symptom Rating Scale (GSRS) from baseline to Day 14 of Gluten Challenge; Test type: Other; p = 0.012, t-test, 2 sided
Statistical Analysis 3: Comparison: Day -14 Low Gluten Dose Group vs Day -14 High Gluten Dose Group vs Day 0 Low Gluten Dose Group vs Day 0 High Gluten Dose Group vs Day 3 Low Gluten Dose Group vs Day 3 High Gluten Dose Group vs Day 7 Low Gluten Dose Group vs Day 7 High Gluten Dose Group vs Day 14 Low Gluten Dose Group vs Day 14 High Gluten Dose Group vs Day 28 Low Gluten Dose Group vs Day 28 High Gluten Dose Group; P Value for Gastrointestinal Symptom Rating Scale (GSRS) between high gluten group and low gluten group across study; Test type: Superiority; p = 0.090, ANOVA

ADVERSE EVENTS:
Time Frame: 4 weeks after participant received first dose
Arm/Group | Low Gluten Group | High Gluten Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Gluten Group (N=10) | High Gluten Group (N=10)
Nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant developed heartburn and vomiting after drinking the lactulose/mannitol solution as part of the intestinal permeability test. Patient recovered without intervention.

LIMITATIONS AND CAVEATS:
This study did have few limitations. First, the study was only moderate in size and drawn from a single center. Many subjects had significant inflammation on duodenal biopsy at baseline which may have limited the effect of gluten challenge. Finally, the high and low gluten groups were significantly different in a few factors including time since diagnosis, time on a gluten-free diet and GSRS score.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No